CLINICAL TRIAL: NCT01234987
Title: Diagnosis of Cancer Using Breath Samples
Status: Completed | Type: Observational
Sponsor: Technion, Israel Institute of Technology (Other)
Collaborators: Rambam Hospital (Unknown)
Other Study IDs: DCHHSGCTIL
Record Dates: First submitted 2010-11-03; First posted 2010-11-04 (Estimated); Last update posted 2011-10-28 (Estimated); Status verified 2010-12

CONDITIONS: Cancer
Keywords: Cancer; Breast Cancer; Colon cancer; Lung Cancer
MeSH Terms: conditions — Neoplasms; Breast Neoplasms; Colonic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (3):
- Breast cancer
- Colon cancer
- Lung Cancer

SUMMARY:
The purpose of this study is to collect breath samples from healthy and cancer sick patients. The breath, collected to special bags, will be transferred to laboratories in the Technion and analyzed using an electronic nose system developed in Hossam Haick's labs (Chemical Engineering, Technion). The hypothesis is that based on the analysis of the chemical bio-markers present in the exhaled breath, cancer states can be distinguished from healthy subjects or before and after treatment, allowing a technique for diagnosis of cancer and/or cancer treatment.

ELIGIBILITY:
Inclusion Criteria:

* The cancer is local or homeostatic
* The subject did not undergo surgery for tumor removal, chemotherapy or radiation treatment prior to first sampling
* The subject signed an informed consent form

Exclusion Criteria:

* The subject is addicted to drugs or alcohol
* The subject smoked in the last hour
* There are communication problems with the subject

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People that undergo screening for breast, colon or lung cancers people diagnosed with breast, colon or lung cancers
Sampling Method: Non-Probability Sample

CONTACTS AND LOCATIONS:
Locations (1):
- Rambam Health Care Campus, Haifa, Israel